CLINICAL TRIAL: NCT04658459
Title: Proximal Interphalangeal Joint Arthroplasty With the TACTYS® Prosthesis : Clinical and Radiographic Results at Medium Term.
Brief Title: Results of the Tactys Implant in Proximal Interphalangeal Joint Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI110
Record Dates: First submitted 2020-11-17; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-11

CONDITIONS: Interphalangeal; Osteoarthritis, Proximal (Bouchard)
Keywords: tactys prosthesis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Results at short term follow up: Functional and Radiological results at short-term follow up (one year at least)
  Interventions: Procedure: Proximal Interphalangeal Joint Arthroplasty with the Tactys Prosthesis
- Results at middle term follow up: Functional and Radiological results at the last follow up of the patient (2 years at least)
  Interventions: Procedure: Proximal Interphalangeal Joint Arthroplasty with the Tactys Prosthesis

INTERVENTIONS:
Procedure: Proximal Interphalangeal Joint Arthroplasty with the Tactys Prosthesis

SUMMARY:
Study at middle term of the functional and radiographic results of proximal interphalangeal joint arthroplasty with the Tactys prothesis. The aim is to evaluate if the short term results are maintained in time.

DETAILED DESCRIPTION:
The inclusion criteria is any patient who has undergone a proximal interphalangeal joint arthroplasty with the Tactys prothesis between january 2015 to january 2020 in the Centre Chirurgical Emile Gallé in Nancy.

The functional results evaluated are range of motion, force, pain, functional score as Quick DASH and the radiological one are clinodactyly, periprosthetic ossifications and loosening, dislocation and implant subsidence.

Data is registered from the medical folder of every patient.

ELIGIBILITY:
Inclusion Criteria:

* one or more proximal interphalangeal joint arthroplasty of long fingers with the Tactys prosthesis
* between january 2015 to january 2020
* major
* centre chirurgical emile gallé, centre hospitalier régional universitaire de Nancy

Exclusion Criteria:

* minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have undergone a proximal interphalangeal joint arthroplasty with the Tactys prosthesis between january 2015 and january 2020 in the Chirugie de la main service in the Centre chirurgical Emile Gallé in Nancy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
range of motion in degrees | minimal one year post-operative
  measurement of range of motion in degrees
force in kilograms | minimal one year post-operative
  measurement of force with jamar and pinch tests in kilograms
pain with the digital pain scale | minimal one year post-operative
  measurement of pain with the digital pain scale to zero to ten
functional score with the Quick DASH | minimal one year post-operative
  measurement of the quick-DASH functional score to zeo to hundred

SECONDARY OUTCOMES:
register the complication and their apparition in time | minimal one year post-operative
assess satisfaction | minimal one year post-operative
  assess the patient's satisfaction : very satisfied, satisfied, moderate, not satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire, Nancy, Meurthe ET Moselle, France